CLINICAL TRIAL: NCT03378882
Title: Research for Angiostrongylus Cantonensis and Costaricensis in French West Indies and French Guiana: a Clinical and Environmental Study
Brief Title: Research for Angiostrongylus Cantonensis and Costaricensis in French West Indies and French Guiana
Acronym: ACCRAG
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Center of Martinique (Other)
Collaborators: University Hospital Center of Pointe-à-Pitre/Abymes (Guadeloupe) (Unknown); Hospital Center of Basse-Terre (Guadeloupe) (Unknown); Hospital Center of Cayenne (French Guiana) (Unknown); Hospital Center of Saint-Laurent du Maroni (French Guiana) (Unknown)
Responsible Party: Sponsor
Other Study IDs: 17/E/05
Record Dates: First submitted 2017-12-07; First posted 2017-12-20 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-12

CONDITIONS: Angiostrongylosis; Hypereosinophilia
Keywords: Angiostrongylosis; Hypereosinophilia; Eosinophilic meningitis; Meningoencephalitis; Achatina fulica; Angiostrongylus cantonensis; Angiostrongylus costaricensis
MeSH Terms: conditions — Strongylida Infections; Eosinophilia; Meningoencephalitis; Angiostrongyliasis | interventions — Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Parasitic serologies — Suspected angiostrongylosis - Angiostrongylus cantonensis:
  * An aliquot of CSF and an aliquot of serum will be sent to the laboratory of tropical medicine in Switzerland for research of specific antibodies.
  * A CSF aliquot will be sent to the CDC for PCR.
  Suspected angiostrongylosis- Angiostrongylus costaricensis:
  - An aliquot of serum will be sent to the laboratory of tropical medicine in Switzerland for research of specific antibodies.
Procedure: Biopsy — Suspected angiostrongylosis - Angiostrongylus costaricensis:
  - A piece of biopsy or intestinal resection will be sent to the pathology laboratory for parasitic elements suggestive of Angiostrongylus costaricensis infection

SUMMARY:
Hospitals in the French West Indies (Fort-de-France (Martinique); Basse-Terre and Pointe-à-Pitre (Guadeloupe); and French Guiana (Cayenne, Saint-Laurent du Maroni)) have noted the emergence of eosinophilic meningitis cases in recent years. This finding is part os eosinophilic meningitis cases emergence and meningoencephalitis caused by the parasite Angiostrongylus cantonensis on the American continent and in the Greater Antilles.

In 2013, the investigation of an eosinophilic meningitis case by the Basse-Terre hospital team with a positive specific PCR in the CSF (CDC, Atlanta, USA) showed the first case of neuromeningeal angiostrongylosis in Guadeloupe. A similar case was diagnosed by serology at Pointe-à-Pitre University Hospital a few years earlier without having been published, and another serious case diagnosed also at Pointe-à-Pitre University Hospital Center in January 2017. The team at the Martinique University Hospital Center also reported several cases of eosinophilic meningitis with positive serologies for A. cantonensis carried out in laboratories outside Martinique (Laboratory of Parasitology, Gonesse, France; Thailand; and Tropical Institute and Public Health, Switzerland) in recent years.

The emergence of this parasitosis is related to the introduction of the intermediate host Achatina fulica on the American continent and the geographical evolution of the angiostrongylosis cases is intrinsically linked to that of the Achatins. To date, only two studies report the environmental presence of Angiostrongylus cantonensis in the Lesser Antilles. One proved the presence in rats (23.4%) on the island of Grenada, and the other in Guadeloupe, showing that 32.4% of Achatina fulica collected carried the parasite by specific PCR. In Martinique, where the number of cases is increasing, and in French Guiana, where there is an increase in the number of cases in neighboring countries, especially Brazil, no study has been conducted on this parasite.

In parallel with this finding, several serious digestive tables associated with strong hypereosinophilia were reported in Martinique and Guadeloupe in the 90s but also in recent years, the last case in December 2016. Etiological diagnoses were established by the discovery of Angiostrongylus costaricensis parasite in ileal pathological specimens. However, these cases could never be investigated by serology or specific PCR due to lack of diagnostic tools available in the French West Indies and Guiana region, and more broadly in metropolitan France.

DETAILED DESCRIPTION:
Angiostrongylosis is a parasitosis caused by the nematode Angiostrongylus sp. The adult parasite lives in the rat's arteries (Rattus norvegicus and Rattus rattus), its definitive host, where it breeds. Stage 1 immature larvae are released into the environment in rat droppings. Stage 3 larval maturation, which is essential for the re-contamination of final hosts, is mainly carried out in the Buyina fulica mollusc (common name: Achatine).

The mode of contamination in humans is by ingestion of stage 3 parasitic larvae according to various modes: accidental ingestion of molluscs or salads soiled by "molluscan slime" (example: by consumption of salad, vegetables, non-washed fruits), voluntary ingestion of molluscs, manipulation of molluscs (children or fishermen), use of drinking water drawn from natural and non-disinfected water bodies. Hand-carried transmission after handling of Achatines is most often reported in young children.

In humans, these larvae have a different preferential tropism depending on the species of Angiostrongylus. The two main pathogenic species for humans are Angiostrongylus cantonensis and Angiostrongylus costaricensis.

Angiostrongylus cantonensis:

After ingestion by man, the larvae of Angiostrongylus cantonensis migrate to the central nervous system. They cause eosinophilic angiostrongyl meningitis and meningoencephalitis, which can lead to severe neurological sequelae (paralysis) or even death.

These clinical features are associated with eosinophilic pleocytosis in CSF (eosinophilic meningitis) and blood eosinophilia.

Angiostrongylus cantonensis was first described in Canton, China in 1935. To date, it is present in the Pacific Islands, Australia, Africa and recently on the American continent.

Angiostrongylus costaricensis:

After ingestion, the larvae of Angiostrongylus costaricensis migrate intestines and into the abdominal cavity. They cause severe abdominal pain mimicking those of appendicitis, haemorrhage and perforation digestive that can lead to death (2 to 8% of cases).

A major eosinophilia usually accompanies these unspecific clinical pictures. Angiostrongylus costaricensis does not have the same geographical distribution as Angiostrongylus cantonensis. It was first described in Costa Rica in 1967 and is endemic on the American continent, where it is at the origin of many human cases.

ELIGIBILITY:
Inclusion Criteria:

* Hypereosinophilia associated with a meningeal table (= suspicion of neuromeningeal angiostrongylosis), or,
* Hypereosinophilia associated with a severe gastrointestinal table(= suspicion of intestinal angiostrongylosis)

Exclusion Criteria:

* Refusal of the patient to be included in the study
* Angiostrongylosis of importation (contracted outside the French West Indies - French Guiana region)
* Absence of hypereosinophilia
* Hypereosinophilia in the context of an other parasitosis
* Non-parasitic hypereosinophilia

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All hospitalized patients, whatever their age, sex, weight, presenting hypereosinophilia.
  Suspicious cases may come from different hospital services (pediatrics, infectiology, resuscitation, neurology, emergencies, ...).
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2018-04-03 (Actual); Primary Completion 2021-04-03 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with angiostrongylosis A. cantonensis | 36 months
  The crude incidence will be calculated: Reported number of cases of angiostrongylosis A. cantonensis diagnosed during the study inclusion period (3 years) on the total population (population census data).
  The number of human cases of angiostrongylosis A. cantonensis diagnosed since the emergence of the parasite in the West Indies and Guiana will be calculated.
  The standardized incidence (on age and sex) of this infection will be calculated.
Number of participants with angiostrongylosis A. costaricensis | 36 months
  The crude incidence will be calculated: Reported number of cases of angiostrongylosis A. costaricensis diagnosed during the study inclusion period (3 years) on the total population (population census data).
  The number of human cases of angiostrongylosis A. costaricensis diagnosed since the emergence of the parasite in the West Indies and Guiana will be calculated.
  The standardized incidence (on age and sex) of this infection will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole DESBOIS, MD, Principal Investigator — CHU of Martinique
Locations (1):
- CHU of Martinique, Fort-de-France, France

IPD SHARING:
Plan to Share IPD: No